CLINICAL TRIAL: NCT04343066
Title: Clinical and Radiographic Evaluation of Bone Remodeling Around Implants With Two Different Surfaces Placed in Horizontally Augmented Bone: a 1-year Randomized Controlled Study
Brief Title: Bone Remodeling Around Implants With Two Different Surfaces Placed in Horizontally Augmented Bone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Nada BOU ABBOUD NAAMAN, Full Professor, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMD195
Record Dates: First submitted 2020-04-03; First posted 2020-04-13 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Dental Implantation; Bone Remodeling
Keywords: Alveolar ridge augmentation; Dental implants; Marginal bone remodeling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- External hex implant (Experimental): External hexagone implant connection
  Interventions: Device: Implant insertion
- Internal hex implant (Experimental): Internal implant connection
  Interventions: Device: Implant insertion

INTERVENTIONS:
Device: Implant insertion — In both groups, the implants will be placed using a two-stage surgical approach at the crestal level in previously horizontally augmented bony sites.
  A final crown will be placed (screw-retained on multiunit abutment) between 3- and 4-months post-implant placement.
  Random allocation of implant type per site will be done by the sealed envelope method.
  Follow-up measurements will be done at 6 months and 1-year post-loading. The measurements are done by a blinded investigator. Before starting the study, the examiner will be trained in a calibration process.
  Exam sheets are kept confidential and anonymous. Inclusion criteria are: patient aged 20 to 65, no systematic contraindication for implant surgery, smoking < 10 cigarettes, previous horizontal bone augmentation, FMBS <20% and FMPS < 20%. Exclusion criteria are: general contraindication for implant surgery, pregnant/lactating women, uncontrolled diabetics, patients not willing to sign the consent form, active periodontitis.
  Other Names: Radiological bone level

SUMMARY:
The aim of this prospective controlled clinical trial is to evaluate the clinical and radiographical outcomes of two implant surfaces inserted in a crest that has been horizontally augmented at least 6 months prior to the implant placement. The horizontal GBR should be done with a xenogenic graft mixed with autologous bone particles, and a collagen membrane stabilized using tacks or screws.

DETAILED DESCRIPTION:
This is a prospective, randomized clinical and radiographical evaluation of bone remodeling around implants with two different surfaces placed in a previously augmented crest.

Patients requiring dental implants in previously horizontally augmented bone crest are recruited at the Department of Periodon¬tics, Faculty of dental medicine, Saint-Joseph University, Beirut, and will be treated with either T3 (contemporary hybrid collar), tapered, ex-hex, CP4 or Full Osseotite, tapered, ex-hex, CP4.

A total of 30 implants will be placed (15 per group). Random allocation of implant type per site will be done by the sealed envelope method.

The implants will be placed using a one-stage surgical approach. A final crown will be placed (screw-retained on multiunit abutment) between 3 and 4 months post-implant placement.

The patients will be followed-up at 6 months and 1 year. Only patients meeting inclusion/exclusion criteria and providing a dated and signed informed consent form will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient age: between 20 and 65
* No systematic contraindication for implant surgery
* No more than 10 cigarettes/day
* Previous horizontal bone augmentation 6 months prior to implant placement
* Adequate oral hygiene i.e. Full mouth bleeding score (FMBS) <20% and Full mouth plaque score (FMPS) < 20%)

Exclusion Criteria:

* Smokers more than 10 cigarettes/day
* Pregnant/lactating women
* Alcoholics/drug addicts
* Uncontrolled diabetics, immunocompromised, blood hemostasis problems
* Patients taking IV bisphosphonates or drugs affecting bone metabolism or mucosal healing
* Patients not willing to sign the consent form
* History of radiotherapy in the head and neck region in the last 5 years
* Active periodontitis on the remaining teeth

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of alveolar ridge thickness at 4 months | During procedure and at 4 months
  Peroperative surgical measurements of the alveolar ridge width at implant sites
Change from baseline of radiographic bone level on CBCT at 1 year post-op | During procedure and at 1 year
  CBCT for buccal bone thickness measurements of the bone crest width at the implant site.
Change from baseline of radiographic bone level assessment at 1 year post-op, on periapical x-ray | During procedure, at 4 months, at 6 months and 1 year
  Radiographic measurements on standardized periapical radiograph of the bone dimensions, for interproximal bone remodeling, from the shoulder of the implant (reference point), to the coronal bone to implant contact
Change from baseline of bone plate thickness at 4 months | During procedure and at 4 months
  Peroperative buccal and lingual residual bone thickness following implant insertion

SECONDARY OUTCOMES:
Insertion torque | During procedure
  Manual torque insertion are registered at implant placement.
Change of Clinical parameters from baseline to 1 year post-op | During procedure, at 6 months and at 1 year
  FMBS, FMPS,
Change of FMBS parameters from baseline to 1 year post-op | During procedure, at 6 months and at 1 year
  Change in full mouth bleeding score
Change of Keratinized tissue height from Baseline to 4 months | During procedure and at 4 months
  Measured using a 1.0-mm marked periodontal probe
Histological analysis | During procedure
  Bone core taken with a 2mm trephine bur at the site of implant placement for non-demineralized histological assessment of regenerated bone quality
Change of FMPS parameters from baseline to 1 year post-op | During procedure, at 6 months and at 1 year
  Change in full mouth plaque score

CONTACTS AND LOCATIONS:
Overall Officials: Nada Naaman, PhD, Principal Investigator — Saint-Joseph University
Locations (1):
- Saint-Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
The outcome measurements and patients characteristics might be shared
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1 year from date of publication
Access Criteria: Following a direct request, for meta-analysis or literature review report.

REFERENCES:
- [Background] Shi JY, Jie-Ni, Zhuang LF, Zhang XM, Fan LF, Lai HC. Peri-implant conditions and marginal bone loss around cemented and screw-retained single implant crowns in posterior regions: A retrospective cohort study with up to 4 years follow-up. PLoS One. 2018 Feb 5;13(2):e0191717. doi: 10.1371/journal.pone.0191717. eCollection 2018. PMID 29401469
- [Background] Liu J, Kerns DG. Mechanisms of guided bone regeneration: a review. Open Dent J. 2014 May 16;8:56-65. doi: 10.2174/1874210601408010056. eCollection 2014. PMID 24894890
- [Background] Koller CD, Pereira-Cenci T, Boscato N. Parameters Associated with Marginal Bone Loss around Implant after Prosthetic Loading. Braz Dent J. 2016 May-Jun;27(3):292-7. doi: 10.1590/0103-6440201600874. PMID 27224562
- [Background] Wennerberg A, Hallgren C, Johansson C, Danelli S. A histomorphometric evaluation of screw-shaped implants each prepared with two surface roughnesses. Clin Oral Implants Res. 1998 Feb;9(1):11-9. doi: 10.1034/j.1600-0501.1998.090102.x. PMID 9590940
- [Background] Rosa MB, Albrektsson T, Francischone CE, Schwartz Filho HO, Wennerberg A. The influence of surface treatment on the implant roughness pattern. J Appl Oral Sci. 2012 Sep-Oct;20(5):550-5. doi: 10.1590/s1678-77572012000500010. PMID 23138742
- [Background] Esposito M, Ardebili Y, Worthington HV. Interventions for replacing missing teeth: different types of dental implants. Cochrane Database Syst Rev. 2014 Jul 22;(7):CD003815. doi: 10.1002/14651858.CD003815.pub4. PMID 25048469
- [Background] Donati M, Ekestubbe A, Lindhe J, Wennstrom JL. Marginal bone loss at implants with different surface characteristics - A 20-year follow-up of a randomized controlled clinical trial. Clin Oral Implants Res. 2018 May;29(5):480-487. doi: 10.1111/clr.13145. Epub 2018 Mar 23. PMID 29569767
- [Background] Testori T, Wiseman L, Woolfe S, Porter SS. A prospective multicenter clinical study of the Osseotite implant: four-year interim report. Int J Oral Maxillofac Implants. 2001 Mar-Apr;16(2):193-200. PMID 11324207
- [Background] Zetterqvist L, Feldman S, Rotter B, Vincenzi G, Wennstrom JL, Chierico A, Stach RM, Kenealy JN. A prospective, multicenter, randomized-controlled 5-year study of hybrid and fully etched implants for the incidence of peri-implantitis. J Periodontol. 2010 Apr;81(4):493-501. doi: 10.1902/jop.2009.090492. PMID 20367092
- [Background] Nevins M, Mellonig JT, Clem DS 3rd, Reiser GM, Buser DA. Implants in regenerated bone: long-term survival. Int J Periodontics Restorative Dent. 1998 Feb;18(1):34-45. PMID 9558555